CLINICAL TRIAL: NCT02543632
Title: PARACHUTE V: PercutAneous Ventricular RestorAtion in Chronic Heart FailUre Due to Ischemic HearT DiseasE. A German Trial to Evaluate the Improvement in Quality of Life and Cardiac Output Following Implanting of the Parachute Implant System
Brief Title: PARACHUTE V PercutAneous Ventricular RestorAtion in Chronic Heart FailUre Due to Ischemic HearT DiseasE.
Acronym: P5
Status: Terminated | Type: Observational
Why Stopped: Company closed
Sponsor: CardioKinetix, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RD1591
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure; Left Ventricular Dysfunction
Keywords: heart failure; parachute; partitioning device
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated group: Subjects who meet the inclusion/exclusion criteria listed and also are approved via anatomical inclusion criteria for treatment with the Parachute Implant System.
  Interventions: Device: Parachute Implant System
- Control group: Subjects who meet the inclusion/exclusion criteria listed and also are are excluded for treatment with the Parachute Implant System due to anatomical characteristics such as obstructing pseudochordae, calcification, or wall thickness.

INTERVENTIONS:
Device: Parachute Implant System — The CardioKinetix Parachute Implant partitions an enlarged ventricle into dynamic and static chambers. The static chamber is a portion of the left ventricular volume that is taken out of circulation. Stresses placed on the partitioned myocardium and the forces transmitted to the apical segment are decreased both in diastole and systole, eliminating the forces responsible for left ventricular dilation. In addition to this regional unloading, the reduction in size of the dynamic chamber results in a decrease of the myocardial stress in the normal myocardium via Laplace Law, providing a global unloading of the ventricle.
  Other Names: Parachute Device
  Groups: Treated group

SUMMARY:
Prospective, multi-center, post-market, non-randomized, nested-control, observational study of the CE marked CardioKinetix Parachute Implant System.

DETAILED DESCRIPTION:
Prospective, multi-center, post-market, non-randomized, nested-control, observational study of the European Conformity Approved (CE marked) CardioKinetix Parachute Implant System. The primary objective is to establish quality-of-life and cardiac output benefit of the Parachute Implant of patients presenting with symptoms of heart failure due to ischemic heart disease. A maximum of 105 treated patients and approximately 25 control patients may be enrolled, with a maximum of 25 treated patients enrolled from any one center. The Primary Endpoint is an improvement of Quality of Life of patients treated with the Parachute Implant at 6 months compared to baseline using the Minnesota Living with Heart Failure (MLWHF) Questionnaire. The Secondary Endpoint is an improvement in Stroke Volume Index (mL/m2) of patients treated with the Parachute Implant at post-procedure compared to pre-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Post MI structural heart dysfunction represented by left ventricular (LV) wall motion abnormality (WMA)
* Symptomatic Heart Failure with reduced Ejection Fraction (EF) (≤ 40%)
* Receiving stable medication for heart failure according to the European Society of Cardiology (ESC) Heart Failure (HF) Guidelines
* >18 years of age
* Provide written informed consent
* Agree to the protocol-required follow-up

Exclusion Criteria:

* Acute myocardial infarction (MI) of the left anterior descending territory within 90 days of enrollment or patients with suspected evolving MI at time of enrollment
* Cardiogenic shock within 72 hours of enrollment
* A known hypersensitivity or contraindication to aspirin, warfarin, nitinol (titanium and nickel alloy), or sensitivity to contrast media, which cannot be adequately pre medicated
* Other hemodynamically structural heart interventions or heart failure device treatment at time of Parachute implant, e.g. mitral valve clip or cardiac resynchronization therapy).
* Co-morbidities associated with a life expectancy of less than 12-months
* Treatment Arm only (Control Arm excluded from this criteria): Anatomical characteristics not suitable for treatment with the Parachute Implant device as screened by magnetic resonance imaging (MRI) or computerized tomography (CT). (Characteristics include inappropriate size and shape of the left ventricle, pseudo chordae or trabeculations interfering with device placement.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age with symptoms of heart failure and anteroapical wall motion abnormality due to myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  An improvement of Quality of Life of patients treated with the Parachute Implant at 6 months compared to baseline (day -1) using the Minnesota Living with Heart Failure (MLWHF) Questionnaire.

SECONDARY OUTCOMES:
Stroke Volume Index | 0 days (at implant)
  An improvement in Stroke Volume Index (mL/m2) of patients treated with the Parachute Implant at post-procedure compared to pre-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Helge Möllmann, MD, Principal Investigator — Kerckhoff Klinik
Locations (10):
- Germany (10):
  - Cardiac Research GmbH, Dortmund, Hohe Straße 1
  - Elisabeth Krankenhaus Essen, Klinik für Kardiologie und Angiologie, Essen, Klara-Kopp-Weg 1
  - Universitätsklinikum Düsseldorf, Klinik für Kardiologie, Pneumologie und Angiologie, Düsseldorf, Moorenstr. 5
  - Uniklinik Aachen, Aachen
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Unfalkrankenhaus Berlin, Berlin
  - University Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Asklepios Klinik St. George, Hamburg
  - Universitäres Herzzentrum Hamburg Eppendorf GmbH, Hamburg